CLINICAL TRIAL: NCT01555398
Title: Open-label, Randomized Study to Evaluate the Effect of Food on the Pharmacokinetic Characteristics of Fenofibric Acid for HIP0901 Capsule in Healthy Male Subjects
Brief Title: Clinical Trial to Evaluate the Effect of Food on the Pharmacokinetic Characteristics of HIP0901 Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-FEN-102
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Fenofibric acid; HIP0901; food effect
MeSH Terms: interventions — fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting conditions (Experimental): Investigational product administrated under fasting condition.
  Interventions: Dietary Supplement: HIP0901 capsule (Fenofibric acid) Fasting conditions/ Fed conditions
- Fed conditions (Active Comparator): Investigational product administrated 30min after starting a high-fat breakfast.
  Interventions: Dietary Supplement: HIP0901 capsule (Fenofibric acid) Fasting conditions/ Fed conditions

INTERVENTIONS:
Dietary Supplement: HIP0901 capsule (Fenofibric acid) Fasting conditions/ Fed conditions — The study drug(HIP0901 capsule(Fenofibric acid, 135mg)) will be administrated under fed or fasting conditions

SUMMARY:
The purpose of this study is to evaluate the effect of food on the pharmacokinetic characteristics of fenofibric acid for HIP0901 capsule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age between 20 and 45
* Informed of the investigational nature of this study and voluntarily agree to participate in this study
* Weight>50kg, BMI of >18kg/m2 and <27kg/m2 subject

Exclusion Criteria:

* Acute disease within 28 days prior to start of study drug administration
* Use of any prescription medication within 14 days prior to Day 1
* Use of any medication within 7 days prior to Day 1
* Has a severe medical history of hypersensitivity to fibric acid derivative
* Participation in another clinical study within 30 days prior to start of study drug administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
AUC of Fenofibric acid | 0-96 hrs
Cmax of Fenofibric acid | 0-96 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea